CLINICAL TRIAL: NCT06391541
Title: Comparison of the Effects of Modified Thoracolumbar Interfacial Plan Block (mTLIP) and Intertransverse Process Block in Lumbar Disc Surgery
Brief Title: mTLIP vs. ITP Blocks in Lumbar Disc Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Çağdaş Baytar, Principal Investigator, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2024/06-18
Record Dates: First submitted 2024-04-26; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Lumbar Disc Herniation; Pain, Postoperative; Regional Aneshesia
Keywords: postoperative pain; opioid consumption; Pain management; nerve blocks; QoR-15
MeSH Terms: conditions — Intervertebral Disc Displacement; Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Control (No Intervention)
- Group mTLIP (Active Comparator)
  Interventions: Procedure: modified thoracolumbar interfacial plan block (mTLIP)
- Group ITP (Active Comparator)
  Interventions: Procedure: Intertransverse process block (ITP)

INTERVENTIONS:
Procedure: modified thoracolumbar interfacial plan block (mTLIP) — Injecting local anesthetic at L3 vertebral level between the longisimus and iliocostalis muscles within the erector spinae muscles.
  Arms: Group mTLIP
Procedure: Intertransverse process block (ITP) — injection of local anesthetic on the superior costotransverse ligament between the transverse process and the pleura.
  Arms: Group ITP

SUMMARY:
to compare ultrasonography (USG)-guided intertransverse process block and modified thoracolumbar interfascial plan (mTLIP) block in the treatment of postoperative pain in patients undergoing lumbar disc herniation surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old
* ASA I-II-III risk group
* Patients whose consent was obtained with an informed consent form
* Patients who will undergo lumbar disc herniation surgery

Exclusion Criteria:

* Patients who refused to participate in the study
* Allergic to local anesthetics
* Patients with coagulopathy
* Infection at the site of intervention
* Patients under 18 years of age
* Patients with ASA score IV and above
* Chronic pain disorders
* Those with neurological or neuromuscular disease
* Patients with psychiatric problems
* Patients with a history of opioid use
* Chronic use of NSAIDs
* Those contraindicated for regional anesthesia
* Patients with a history of opioid use
* Chronic analgesic use

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
postoperative opioid consumption | up to 24 hours after surgery
  total amount of opioids consumed in 24 hours postoperatively

SECONDARY OUTCOMES:
pain scores | up to 24 hours after surgery
  Patients will be evaluated at regular intervals after surgery and their pain will be measured using a numerical rating scale.
incidence of nausea and vomiting | up to 24 hours after surgery
  nausea and vomiting of postoperative patients will be evaluated
Quality of Recovery-15 scale | 24 hours after surgery
  The quality of recovery of patients will be assessed with the quality of recovery 15 questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University medicine faculty, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No